CLINICAL TRIAL: NCT01210612
Title: The Effect of Five-Toed Socks on Postural Control Among Active Individuals Who Have Chronic Ankle Instabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Phillip Gribble, Principal Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UTHSC-12
Record Dates: First submitted 2010-06-23; First posted 2010-09-28 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without Unilateral CAI (Active Comparator): Individuals with no history of chronic ankle instability (CAI)
  Interventions: Device: Unilateral CAI
- With Unilateral CAI (Experimental): Individuals with a history of chronic ankle instability (CAI) that is affecting only one limb
  Interventions: Device: Unilateral CAI

INTERVENTIONS:
Device: Unilateral CAI — five-toed socks usage

SUMMARY:
Lateral ankle sprain (LAS) is one of the most common injuries in sports. There is a unique style of socks that have become popular in Japan among athletes that could also improve postural control. The purpose of the study is to determine the effectiveness of five-toed socks on dynamic postural control in individuals with and without chronic ankle instability.

DETAILED DESCRIPTION:
Lateral ankle sprain (LAS) is one of the most common injuries in sports. Ankle braces and orthotic insoles also have been shown to influence the neuromuscular control system by enhancing the proprioceptive and cutaneous afferent inputs to the central nerve system; thereby improving postural control. There is a unique style of socks that have become popular in Japan among athletes that could also improve postural control by enhancing cutaneous afferent inputs from the plantar surface of the foot and toes. The purpose of the study is to determine the effectiveness of five-toed socks on dynamic postural control in individuals with and without chronic ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* member of university community
* All subjects will be physically active (at least 30 minutes of sustained exercise 3 times/week

Exclusion Criteria:

* history of: knee or hip musculoskeletal injury or surgery
* history of: fracture or dislocation of the testing ankle or leg
* neurological problems
* vestibular disorders or concussions within the last 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Gribble, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period was from January 2009 to September 2010. Data was collected at Athletic Training Research Laboratory located in room 1406A Health Science and Human Service Building, University of Toledo, Toledo, OH 43606. Subjects were approached in groups during classes at the University of Toledo.
Pre-assignment Details: Enrolled participants were selected based on the inclusion and exclusion criteria in this study, therefore no participants were excluded following participant enrollment, but prior to group assignment.
Groups:
- With Unilateral CAI; Without Unilateral CAI: five-toed socks : five-toed socks usage
Period: Overall Study
Arm/Group | With Unilateral CAI | Without Unilateral CAI
Started | 23 | 30
Completed | 23 | 28
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | With Unilateral CAI | Without Unilateral CAI | Total
Number analyzed (Participants) | 23 | 30 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 30 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (3.3) | 22.7 (3.0) | 22.5 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 16 | 21 | 37
Region of Enrollment [Number; unit: participants]
  United States | 23 | 30 | 53

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measurement for This Study Was to Determine Differences in Center of Pressure (COP) and Static Postural Control Patterns in Individuals With and Without CAI During the Single Limb Balance Test.
Description: Participants were recruited to complete three testing sessions, separated by approximately one week. The participants were tested while wearing five-toed socks. Static postural control was assessed on a force plate (model 4060NC; Bertec Corp. Inc., Columbus, OH) with the subject in a single-limb stance. Center of Pressure (COP) data were sampled at 50Hz. The subjects completed three 15-second trials with a one-minute rest between trials. Motion Monitor software (Innovative Sports Training, Inc., Chicago, IL) collected COP data during the single-limb stance test. The primary outcome was COP-Velocity (cm/sec).
Time Frame: 3 weeks
Population: In published data by the lab director in which the dependant variable was normalized reaching distance on the SEBT, CAI subjects experienced a significantly reduced anterior reaching direction on their injured side compared to the Control group. Based on these data, to achieve a power level of 0.80, fifteen subjects in each group will be needed.
Measure: Mean (Standard Deviation); unit: COP-Velocity (cm/sec)
Groups:
- With Unilateral CAI: Participants with unilateral CAI while wearing five-toed socks
- Without Unilateral CAI: Participants without unilateral CAI while wearing five-toed socks
Arm/Group | With Unilateral CAI | Without Unilateral CAI
Number analyzed (Participants) | 23 | 28
COP-Velocity (cm/sec)
  Eyes Open | 0.61 (0.27) | 0.55 (0.21)
  Eyes Closed | 1.31 (0.38) | 1.26 (0.34)

2. Secondary Outcome: Reaching Distances
Description: The secondary outcome measurement for this study will be to determine differences in the mean value of the three reaching distances (the anterior, posterior lateral, and posterior medial direction) of the SEBT in individuals with and without chronic ankle instability. The reaching distances (cm) from the three directions were averaged together and then normalized to the leg length of the stance leg (cm). The outcome variable, normalized maximum reaching distance (MAXD), was represented as a percentage value representing the distance as a % of leg length.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: MAXD (% of leg length)
Arm/Group | With Unilateral CAI | Without Unilateral CAI
Number analyzed (Participants) | 23 | 28
MAXD (% of leg length) | 66.1 (6.4) | 71.4 (5.8)

ADVERSE EVENTS:
Arm/Group | With Unilateral CAI | Without Unilateral CAI
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/30
Other Adverse Events (participants affected / at risk) | 0/23 | 0/30

LIMITATIONS AND CAVEATS:
The day-to-day diurnal effect has been recognized as an important factor to consider when measuring postural control. We, however, did not consider day-to-day influences in postural control. This may have influenced the data we have collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes